CLINICAL TRIAL: NCT03538236
Title: Intragastric Balloon in Combination With Lifestyle Intervention vs. Lifestyle Intervention Alone in Obese Patients Having NASH With Significant Fibrosis
Brief Title: Intragastric Balloon With Lifestyle Intervention vs. Lifestyle Intervention in Obese Patients With NASH
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: The study did not recruit any patients.
Sponsor: Johns Hopkins University (Other)
Collaborators: ReShape Lifesciences (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: IRB00115848
Record Dates: First submitted 2018-05-03; First posted 2018-05-29 (Actual); Last update posted 2021-03-30 (Actual); Status verified 2020-11

CONDITIONS: Obesity; NASH - Nonalcoholic Steatohepatitis; Obesity, Morbid
MeSH Terms: conditions — Obesity; Non-alcoholic Fatty Liver Disease; Obesity, Morbid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Lifestyle intervention alone (Active Comparator): All patients included in the study will undergo an evaluation by a nutritionist and will undergo diet and lifestyle intervention.
  Interventions: Behavioral: Lifestyle intervention
- Intragastric balloon with lifestyle (Experimental): Patients who do not reach the 10% weight loss with lifestyle intervention alone after 6 months will be offered to have intragastric balloon insertion for 6 months. Regardless of whether an intragastric balloon is inserted, all patients will continue with the same lifestyle changes described above for another 6 months.
  Interventions: Device: Intragastric balloon; Behavioral: Lifestyle intervention

INTERVENTIONS:
Device: Intragastric balloon — Intragastric balloon insertion will be performed by an endoscopist under monitored anesthesia care. The Intragastric BalIoon (GB) comes as a deflated balloon pre-loaded on a catheter, which is inserted transorally into the proximal gastric body. An endoscope is then inserted alongside the device allowing for direct visualization of the balloon. Once in place, the intragastric balloon will be filled with saline through an external port. The balloon is inserted for 6 months then retrieved endoscopically
  Arms: Intragastric balloon with lifestyle
Behavioral: Lifestyle intervention — All patients included in the study will undergo an evaluation by a nutritionist. All participants will receive recommendations for a diet. Participants will be instructed to keep a daily food diary and will meet with the nutritionist to reinforce the behavior every 12 weeks for 12 months.

SUMMARY:
The primary objective of this study is to assess efficacy of intragastric balloon for weight loss in obese patients who also concurrently have NASH.

DETAILED DESCRIPTION:
Non-alcoholic steatohepatitis (NASH) is a growing and leading etiology of chronic liver disease worldwide resulting in substantial morbidity and mortality.

Given recent data confirming weight loss as an effective treatment strategy for NASH and the recent availability of endoscopic bariatric therapies recently described by the American Society for Gastrointestinal Endoscopy (ASGE) and approved by the Food and Drug Administration (FDA), the investigators seek to primarily study efficacy of intragastric balloon for weight loss in obese patients having NASH. Secondary objective would be to assess whether the use of intragastric balloon combined with lifestyle intervention can improve liver histology in NASH with significant fibrosis over lifestyle intervention alone in a prospective paired study.

ELIGIBILITY:
Inclusion Criteria:

* Patients with BMI 30-35 (obese individuals who qualify for Intragastric Balloon (IGB) as per FDA but who do not qualify for bariatric surgery)
* Patients with NASH defined as presence of steatosis by ultrasound transient elastography with Controlled Attenuation Parameter (CAP) and persistent elevation in liver enzymes without significant history of alcohol consumption (>21 drinks/week in men and >14 drinks/week in women) and with other etiology of chronic liver diseases excluded including medication induced steatosis
* Severe fibrosis F3-F4 on ultrasound elastography

Exclusion Criteria:

* Suspected or biopsy confirmed liver cirrhosis
* Significant ethanol consumption >21 drinks/week in men and >14 drinks/week in women
* Patients with human immunodeficiency virus (HIV)
* Patients on medications associated with steatohepatitis including amiodarone, diltiazem, corticosteroids, methotrexate, tamoxifen, protease inhibitors, and valproate
* Presence of other chronic liver disease including hepatitis B-C, autoimmune hepatitis, alpha 1 antitrypsin deficiency, Wilson's disease, and hemochromatosis
* Pregnant or breast-feeding
* Patients who already have an intragastric balloon
* Patients with Gastroesophageal reflux disease (GERD)
* Patients with previous gastric surgeries, altered gastrointestinal anatomy such as Billroth I, Billroth II, roux-en-y gastrectomy, roux-en-y hepaticojejunostomy, or any restrictive or bypass bariatric surgery
* Presence of inflammatory disorder of the gastrointestinal tract
* Patients with active peptic ulcer disease
* Patients with gastroesophageal varices
* Presence of a large hiatal hernia (grade IV on Hills classification: large hiatal hernia and essentially no fold approximating the endoscope in the retroflexed view and where the lumen of the esophagus is gaping open allowing the squamous epithelium to be seen)
* Structural abnormality in the esophagus or pharynx
* Have major esophageal motility disorders as per the Chicago classification including achalasia, diffuse esophageal spasm, jackhammer esophagus, and Esophagogastric junction (EGJ) outflow obstruction
* Mucosal or submucosal gastric mass that is clinically suspected to be of malignant nature
* Severe clotting or bleeding disorder
* Other medical condition that does not allow for endoscopic procedure
* Severe psychiatric illness
* Unable to participate in routine medical follow-up
* On antiplatelet agents including clopidogrel, ticlopidine, prasugrel, and cangrelor. Aspirin use will be allowed
* On anticoagulants including heparin, warfarin, dabigatran, rivaroxaban, apixaban, and edoxaban

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-03-01 (Estimated); Primary Completion 2022-05-30 (Estimated); Study Completion 2022-05-30 (Estimated)

PRIMARY OUTCOMES:
Weight loss | 1 year
  Weight lost as a percentage of baseline total body weight

SECONDARY OUTCOMES:
Liver fibrosis | 1 year
  Fibrosis stage on ultrasound transient elastography
Liver panel | 1 year
  Biochemical liver panel
Lipid panel | 1 year
  Lipid panel via blood level measurement
Complications | 1 year
  Complications associated with intragastric balloon using severity grading according to the ASGE lexicon
Glucose | 1 year
  Glucose level will be measured by blood test

CONTACTS AND LOCATIONS:
Overall Officials: Vivek Kumbhari, MD, Principal Investigator — Johns Hopkins University